CLINICAL TRIAL: NCT02092896
Title: Treatment With Liraglutide as add-on to Insulin in Type 1 Diabetic Patients. Effects on Glycemic Control and Counterregulation and Cognitive Performance During Hypoglycaemia
Brief Title: Liraglutide as add-on to Insulin in Type 1 Diabetes
Acronym: T1DMLIRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: NNF Center for Basal Metabolic Research, Denmark (Unknown); Hillerod Hospital, Denmark (Other); Danish PhD schools of Molecular Metabolism and Endocrinology (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Christan SS Frandsen, MD, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-002526-67; 2012-002526-67 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Cognitive performance; Hypoglycemia; Insulin; Glucagon-Like Peptide 1; Hypoglycemic Agents; Physiological Effects of Drugs; Pharmacologic Actions; Incretins; Hormones
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Hypoglycemia; Insulin Resistance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo + Insulin + Study 2 (Placebo Comparator): Study 2: Cognitive performance test
  Interventions: Drug: Liraglutide
- Liraglutide + Insulin + Study 2 (Experimental): Study 2: Cognitive performance test
  Interventions: Drug: Placebo
- Liraglutide + Insulin + Study 1 (Experimental): Study 1: Gastric emptying test
  Interventions: Drug: Liraglutide
- Placebo + Insulin + Study 1 (Placebo Comparator): Study 1: Gastric emptying test
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Subjects randomised to 1.2 mg liraglutide treatment or liraglutide placebo will receive 0.6 mg for 1 weeks followed by 1.2 mg for 11 weeks. At baseline and week 12 study 1 is performed.
  Arms: Liraglutide + Insulin + Study 1
Drug: Placebo — Subjects randomised to 1.2 mg liraglutide treatment or liraglutide placebo will receive 0.6 mg for 1 weeks followed by 1.2 mg for 11 weeks. At baseline and week 12 study 1 is performed.
  Arms: Placebo + Insulin + Study 1
Drug: Liraglutide — Subjects randomised to 1.2 mg liraglutide treatment or liraglutide placebo will receive 0.6 mg for 1 weeks followed by 1.2 mg for 11 weeks. At baseline and week 12 study 2 is performed.
  Arms: Placebo + Insulin + Study 2
Drug: Placebo — Subjects randomised to 1.2 mg liraglutide treatment or liraglutide placebo will receive 0.6 mg for 1 weeks followed by 1.2 mg for 11 weeks. At baseline and week 12 study 2 is performed.
  Arms: Liraglutide + Insulin + Study 2

SUMMARY:
The purpose of this study is to:

Part 1:

To investigate how 12 weeks treatment with liraglutide affects glycemic control in poorly controlled patients and how the treatment affects gastric emptying rate during hypoglycemia.

Part 2:

To investigate how 12 weeks treatment of type 1 diabetic patients with liraglutide affects counterregulatory hormones and cognitive performance during hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* BMI: 18-28
* HbA1c ≥ 8 %
* No residual β-cell function (glucagon test with c-peptide < 60 pM)
* Caucasian
* Diagnosed with type 1 diabetes at 5 to 40 years of age (both inclusive).
* Remission phase must be completed
* Female participants must use adequate contraception
* Informed consent

Exclusion Criteria:

* Overt diabetes complications; creatinin > 130 µM, proliferative retinopathy, macroalbuminuria.
* Autonomic neuropathy (RR-variation </=10 beats/min) and/or Orthostatic hypotension (OH).
* Anemia, Hb concentration; female <7.0 mmol/l, male<8.0 mmol/l
* Pregnancy or lactation
* Epilepsy
* Use of antiepileptic medication
* Use of beta blockers
* Previously apoplexy cerebri.
* Any use of benzodiazepine within the last month
* Any use of neuroleptic drugs within the last six months
* Self-perceived hearing loss
* Alcohol or drug abuse
* Allergy to the medication or placebo.
* Treatment with any medication affecting glucose metabolism.
* Any disorder which in the investigators opinion could interfere with the safety and results of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c (glycosylated haemoglobin) | Week 0, week 12
Changes from baseline in EEG and cognitive performances | week 0, week 12
Change from baseline in gastric emptying rate | week 0, week 12

SECONDARY OUTCOMES:
Change from baseline in glycemic control (CGM) | week 0, week 12
Change from baseline in total daily insulin dose | week 0, week 12
Changes from baseline in the counterregulatory hormone responses during hypoglycemia | week 0, week 12
Change from baseline in body weight | week 0, week 12
Change from baseline in auditory evoked potentials (AEP) during hypoglycemia | week 0, week 12
Change from baseline in corrected QTc-interval (QTc) during hypoglycemia | week 0, week 12
Change from baseline in hypoglycemic symptom score | week 0, week 12

OTHER OUTCOMES:
Frequency of Hypoglycemic episodes | Week 0, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Christian SS Frandsen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Dept. of Endocrinology, Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Frandsen CS, Dejgaard TF, Holst JJ, Andersen HU, Thorsteinsson B, Madsbad S. Twelve-Week Treatment With Liraglutide as Add-on to Insulin in Normal-Weight Patients With Poorly Controlled Type 1 Diabetes: A Randomized, Placebo-Controlled, Double-Blind Parallel Study. Diabetes Care. 2015 Dec;38(12):2250-7. doi: 10.2337/dc15-1037. Epub 2015 Oct 20. PMID 26486191